CLINICAL TRIAL: NCT05809115
Title: Neurodevelopmental Outcomes in Children: Strengthening the Caregiver-Child Story
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Episcopal Health Foundation (Unknown)
Responsible Party: Principal Investigator, Michelle Lopez, Associate Professor of Pediatrics, Baylor College of Medicine
Other Study IDs: H-53133
Record Dates: First submitted 2023-03-20; First posted 2023-04-12 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Food Insecurity; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Neurocognitive Outcomes: * Surveys
  * General behavioral, economic, and household resources
- Neurodevelopmental Outcomes: * Surveys
  * Individualized behavioral, economic, and household resources

SUMMARY:
The main goal of this research is to help families who are experiencing food insecurity (FI) and help mothers with depression.

The next goal is to provide other resources to help with household needs like rent or utility assistance, health insurance, anxiety, and depression. Our theory is that helping with food insecurity, household needs, and emotional health will help children and families.

DETAILED DESCRIPTION:
Aim 1: Implement a refined mental health (MH) intervention in caregivers of hospitalized children: sessions with a Behavioral Health Clinician (BHC) with more individualized support based on caregiver-child needs, instruction on caregiver-child bonding, and a streamlined handoff to a community MH provider. Follow-up outcomes include caregiver MH and caregiver-child attachment (survey) and child development (electronic health records, EHR).

Aim 2: Execute an enhanced intervention for FI. All families who screen positive for FI will still receive assistance with public benefit enrollment and access to local food pantries. Families with additional needs will receive support for 10 additional non-medical drivers of health (NMDH). Assistance will be provided by onsite Houston Food Bank (HFB) Community Referral Specialists. Follow-up outcomes include enrollment in public/community resources and food security status (survey).

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of young children (0-36 months of age) hospitalized at Texas Children's Hospital on acute care units.
* English or Spanish speaking caregiver.
* Age of caregiver ≥ 18 years old.
* Hospital day 2 or later of patient admission.

Exclusion Criteria:

* Caregivers who do not have primary custody
* Children in CPS custody
* Caregivers who live outside of Texas (due to lack of Houston Food Bank resources outside of Texas)
* Previous enrollment in this study.
* Patient is in the process of being discharged/observation status administration.
* Caregiver is not the primary caregiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population are the caregivers of children hospitalized at Texas Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Maternal Child Bonding | 6 months
  The validated Maternal Attachment Inventory will be used for data collection. Higher scores indicate greater maternal child bonding.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lopez, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will not be shared with other researchers

REFERENCES:
- [Background] Lopez MA, Yu X, Hetrick R, Raman S, Lee J, Hall J, Tran K, Vonasek B, Garg A, Raphael J, Bocchini C. Social Needs Screening in Hospitalized Pediatric Patients: A Randomized Controlled Trial. Hosp Pediatr. 2023 Feb 1;13(2):95-114. doi: 10.1542/hpeds.2022-006815. PMID 36594231